CLINICAL TRIAL: NCT01940796
Title: Phase I Trial of Brentuximab Vedotin for Refractory Chronic Graft-vs.-Host Disease (GVHD)
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Toxicity
Sponsor: Massachusetts General Hospital (Other)
Collaborators: Seagen Inc. (Industry)
Responsible Party: Principal Investigator, Yi-Bin A. Chen, MD, Principal Investigator, Massachusetts General Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 13-239
Record Dates: First submitted 2013-09-09; First posted 2013-09-12 (Estimated); Last update posted 2018-07-26 (Actual); Status verified 2018-07

CONDITIONS: Graft-vs-Host Disease; GVHD
Keywords: Brentuximab Vedotin; GVHD; Refractory Chronic Graft vs Host Disease
MeSH Terms: conditions — Graft vs Host Disease | interventions — Brentuximab Vedotin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Brentuximab Vedotin (Experimental): The dose of brentuximab Vedotin will be based on the cohort the participant is enrolled on. Dosing will be based on the participant's weight prior to each dose. Actual weight will be used except for participants weighing > 100 kg. The dose for participants weighing > 100 Kg will be calculated based on a weight of 100 kg. The dose should be rounded to the nearest whole number of milligrams. Brentuximab vedotin will be administered over approximately 30 minutes IV.Up to five dose levels will be tested in cohorts of 3-6 participants each. Once the maximum tolerated dose (MTD) is established, 10 more participants will be treated at the MTD for analysis of efficacy.
  Interventions: Drug: Brentuximab Vedotin

INTERVENTIONS:
Drug: Brentuximab Vedotin — Up to five dose levels will be tested in cohorts of 3-6 participants each. Once the maximum tolerated dose (MTD) is established, 10 more participants will be treated at the MTD for analysis of efficacy.

SUMMARY:
This research study is trying to determine the safest dose of Brentuximab Vedotin that can be given to patients with chronic GVHD and see if chronic GVHD improves.

DETAILED DESCRIPTION:
This study is looking for the highest dose of the Brentuximab Vedotin that can be administered safely without severe or unmanageable side effects in patients that have chronic Graft vs. Host Disease, not everyone who participates in this research study will receive the same dose of the study drug. The dose each patient will get depends on the number of participants who have been enrolled in the study prior and how well they have tolerated their doses.

Each patient will receive a dose of Brentuximab Vedotin every 3 weeks. Brentuximab Vedotin is administered via intravenous infusion, or IV infusion, which means directly into the vein, over a period of about 30 minutes.

Each cycle is 21 days long.

Each patient will undergo the following tests and procedures when they come into the clinic to receive each dose of Brentuximab Vedotin:

Days 1, 8, and 15 of 1st 2 cycles:

* Physical exam, which includes height, weight, body surface area and vital signs.
* A medical history, which includes questions about your health, current medications, and any allergies.
* Performance status, which evaluates how participant are able to carry on with your usual activities.
* Routine blood tests to test overall health (about 1 teaspoon of blood) Assessment of side effects- physician will evaluate the patient's current health and ask questions to see there are any experienced side effects from taking the study drug.

Only Day 1 of 1st 3 cycles:

* Research blood draws for biomarker and PK assessments (pharmacokinetic assessments that measure the level of drug in the patient's blood) (about 4 teaspoons of blood)
* Biomarker studies blood draw (about 4 teaspoons) Viral monitoring blood tests to make sure each patient has not developed any new viruses as a result of treatment (about 4 teaspoons of blood)
* Chronic GVHD assessments: The patient's physician may need to perform other tests to confirm the diagnosis of acute GVHD. These can include more blood tests, imaging studies, and possibly biopsies of affected organs. The exact tests will be determined by the patient's physician

Planned Follow-up: If the patient's physician believes the patient is responding well to treatment, the patient may receive up to 16 cycles of Brentuximab Vedotin. The Investigator would like to keep track of patient's medical condition for 12 months after the patient has completed the first 2 cycles of treatment, no matter if the patient receives more doses or not. The Investigator would like to do this by calling the patient on the telephone to see how he/she is doing. Keeping in touch with patient and checking the condition helps the Investigator look at the long-term effects of the research study.

ELIGIBILITY:
Inclusion Criteria:

* Recipients of allogeneic hematopoietic cell transplantation (HCT) after either myeloablative or reduced intensity conditioning regimens. Any donor source of stem cells is eligible.
* Participants must be at least 100 days after HCT.
* Patients must have steroid refractory cGVHD, defined as having persistent signs and symptoms of chronic GVHD (section 13.1) despite the use of prednisone at ≥ 0.25 mg/kg/day (or 0.5 mg/kg every other day) for at least 4 weeks in the preceding 12 months (or equivalent dosing of alternate corticosteroids) without complete resolution of signs and symptoms.
* Stable dose of corticosteroids for 4 weeks prior to enrollment
* No addition or subtraction of other immunosuppressive medications (e.g., calcineurin inhibitors, sirolimus, mycophenolate mofetil) for 4 weeks prior to enrollment. The dose of immunosuppressive medicines may be adjusted based on the therapeutic range of that drug
* Serum Cr ≤ 3 gm / dL
* Adequate hepatic function (total bilirubin < 2.0 mg/dl, AST < 5x ULN), unless hepatic dysfunction is a manifestation of presumed cGVHD. For patients with abnormal LFTs as the sole manifestation of active cGVHD, documented cGVHD on liver biopsy will be required prior to enrollment. Abnormal LFTs in the context of active cGVHD involving other organ systems may also be permitted if the treating physician documents the abnormal LFTs as being consistent with active hepatic cGVHD, and a liver biopsy will not be mandated in this situation.
* Patients must have adequate bone marrow function as defined by ANC ≥ 1000 / µl and platelets ≥ 20,000 / µl without growth factor or transfusional support
* Negative pregnancy test for females of child bearing age
* Age ≥ 18 - The safety and effectiveness of brentuximab vedotin has not been established in the pediatric population. Clinical trials of brentuximab vedotin included only 9 pediatric patients and this number is not sufficient to determine whether they respond differently than adult patients.
* The effects of brentuximab vedotin on the developing human fetus are unknown. For this reason and because chemotherapy agents are known to be teratogenic, women of child-bearing potential and men must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) prior to study entry and for the duration of study participation. Should a woman become pregnant or suspect she is pregnant while participating in this study, she should inform her treating physician immediately.
* Ability to understand and the willingness to sign a written informed consent document

Exclusion Criteria:

* Ongoing prednisone requirement > 1 mg/kg/day (or equivalent)
* Exposure to any new immunosuppressive medication in the 4 weeks prior to enrollment.
* ECP therapy within 4 weeks prior to enrollment
* Active malignant disease relapse
* Active, uncontrolled infection
* Uncontrolled cardiac angina or symptomatic congestive heart failure (NYHA Class III or IV).
* Karnofsky performance status < 30
* Prior use of brentuximab vedotin for GVHD is not allowed. Prior use of brentuximab vedotn for the treatment of malignancy is allowed.
* Pregnant women are excluded from this study because brentuximab vedotin is a chemotherapy agent with the potential for teratogenic or abortifacient effects. Because there is an unknown but potential risk of adverse events in nursing infants secondary to treatment of the mother with brentuximab vedotin, breastfeeding should be discontinued if the mother is treated with brentuximab vedotin.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 19 (Actual)
Dates: Start 2013-10 (Actual); Primary Completion 2016-12 (Actual); Study Completion 2016-12 (Actual)

PRIMARY OUTCOMES:
To define the maximum tolerated dose (MTD) of brentuximab vedotin when given as treatment for refractory chronic GVHD | 2 Years
  To define the maximum tolerated dose (MTD) of brentuximab vedotin when given as treatment for refractory chronic GVHD

SECONDARY OUTCOMES:
To test the overall response rate of Brentuximab Vedotin when given as treatment for refractory chronic GVHD | 2 Years
  To test the overall response rate of Brentuximab Vedotin when given as treatment for refractory chronic GVHD
To identify the toxicities associated with Brentuximab Vedotin when used as therapy for refractory chronic GVHD | 2 Years
  To identify the toxicities associated with Brentuximab Vedotin when used as therapy for refractory chronic GVHD
Overall Survival | 2 Years
  Overall survival at 100 days, 180 days, and one year after first infusion
To assess levels of soluble CD30 and surface CD30 expression on peripheral blood T-cells in participants with chronic GVHD before and after the administration of brentuximab vedotin | 2 Years
  To assess levels of soluble CD30 and surface CD30 expression on peripheral blood T-cells in participants with chronic GVHD before and after the administration of brentuximab vedotin
To assess dose of steroids (mg/kg/day of prednisone equivalent) at 6 and 12 months after starting therapy | 2 Years
  To assess dose of steroids (mg/kg/day of prednisone equivalent) at 6 and 12 months after starting therapy

CONTACTS AND LOCATIONS:
Overall Officials: Yi-Bin Chen, MD, Principal Investigator — Massachusetts General Hospital
Locations (1):
- Massachusetts General Hospital, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Chen YB, Perales MA, Li S, Kempner M, Reynolds C, Brown J, Efebera YA, Devine SM, El-Jawahri A, McAfee SL, Spitzer TR, Soiffer RJ, Ritz J, Cutler C. Phase 1 multicenter trial of brentuximab vedotin for steroid-refractory acute graft-versus-host disease. Blood. 2017 Jun 15;129(24):3256-3261. doi: 10.1182/blood-2017-03-772210. Epub 2017 May 4. PMID 28473406